CLINICAL TRIAL: NCT02410915
Title: Gait Training Early After Stroke - a Comparison Between Training With the Exoskeleton Hybrid Assistive Limb and Conventional Gait Training
Brief Title: A Comparison Between the Exoskeleton Hybrid Assistive Limb and Conventional Gait Training Early After Stroke
Acronym: HAL-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: University of Tsukuba (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Reg. Physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/1807-31/2
Record Dates: First submitted 2015-02-13; First posted 2015-04-08 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Stroke; Gait, Hemiplegic; Ambulation Difficulty; Hemiparesis
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Mobility Limitation; Paresis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Intervention: Hybrid Assistive Limb (HAL); gait training in combination with conventional training. Training with the exosceleton Hybrid Assistive Limb (HAL) is performed in 1 session per day, 4 days per week during 4 weeks. Time for each session is individualised but does not exceed 60 minutes/session (effective time). Training with HAL is performed in combination with body-weight support system and on a treadmill. The training program is performed by 2 physiotherapists, who have been trained in the HAL method.
  Interventions: Device: Hybrid Assistive Limb (HAL); gait training
- Control Group (Active Comparator): Intervention: Conventional gait training is individualized and performed according to current practice (approximately 30-60 minutes/session, 5 days a week) and may include standing, weight shifting, stepping, over ground walking with assistance and/or assistant devices as well as the use of a treadmill and body weight support. Conventional gait training is offered to both study groups.
  Interventions: Other: Control Group; Conventional gait training

INTERVENTIONS:
Device: Hybrid Assistive Limb (HAL); gait training — Training with HAL is performed in 1 session per day, 4 days per week during 4 weeks. Time for each session is individualised but does not exceed 60 minutes/session (effective time). Training with HAL is performed in combination with body-weight support system and on a treadmill. The training program is performed by 2 physiotherapists, who have been trained in the HAL method.
  Other Names: Hybrid Assistive Limb (HAL)
  Arms: Study Group
Other: Control Group; Conventional gait training — Conventional gait training is individualized and performed according to current practice (approximately 30-60 minutes/session, 5 days a week) and may include standing, weight shifting, stepping, over ground walking with assistance and/or assistant devices as well as the use of a treadmill and body weight support. Conventional gait training is offered to both study groups.
  Arms: Control Group

SUMMARY:
Overall aim is to evaluate HAL for gait training early after stroke and the effect of HAL on short- and long-term functioning, disability and health compared to conventional gait training as part of an inpatient rehabilitation program early after stroke.

DETAILED DESCRIPTION:
To compare outcome after 4 weeks of gait training with HAL vs. 4 weeks of conventional gait training as part of a regular inpatient rehabilitation program for hemiparetic patients with severely limited mobility early after stroke.

Study design: Randomized, controlled study with blinded outcome assessment.

Conventional gait training is individualized and performed according to current practice (approximately 30-60 minutes/session, 5 days a week) and may include standing, weight shifting, stepping, over ground walking with assistance and/or assistant devices as well as the use of a treadmill and body weight support. Conventional gait training is offered to both study groups.

Training with HAL is performed in 1 session per day, 4 days per week during 4 weeks. Time for each session is individualised but does not exceed 60 minutes/session (effective time). Training with HAL is performed in combination with body-weight support system and on a treadmill. The training program is performed by 2 physiotherapists, who have been trained in the HAL method.

ELIGIBILITY:
Inclusion Criteria:

* less than 8 weeks since stroke onset; inability to walk independently due to lower extremity paresis (i.e. FAC score 0-1), able to sit on a bench with or-without supervision at least five minutes; sufficient postural control to allow upright position in standing with aids and/or manual support; ability to understand training instructions as well as written and oral study information and to express informed consent; body size compatible with the HAL suit.

Exclusion Criteria:

* contracture restricting gait movements at any lower limb joint; cardiovascular or other somatic condition incompatible with intensive gait training; and severe, contagious infections.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Functional Ambulation Categories (FAC) | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Level of independence in walking, range 0-5

OTHER OUTCOMES:
Change in Gait Deviation Index (GDI) | After 4 weeks of training and 6 months after stroke
  Gait pattern function will be assessed using a motion capture system (Vicon MX40, Oxford, UK) with two force plates (Kistler, Winterthur, Switzerland) and wireless surface electromyography (EMG, Noraxon, Scottsdale, Arizona, USA). Markers will be placed according to a conventional full-body model (Vicon Plug-in-Gait) and surface EMGs, according to standardized electrode placement (www.seniam.org).
Change in GDI-kinetic. | After 4 weeks of training and 6 months after stroke
  Gait pattern function will be assessed using a motion capture system (Vicon MX40, Oxford, UK) with two force plates (Kistler, Winterthur, Switzerland) and wireless surface electromyography (EMG, Noraxon, Scottsdale, Arizona, USA). Markers will be placed according to a conventional full-body model (Vicon Plug-in-Gait) and surface EMGs, according to standardized electrode placement (www.seniam.org).
Change in Barthel Index | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Independence in mobility and personal care
Change in Fugl-Meyer for Lower extremities | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Sensory and motor function in lower extremities
Change in Berg Balance scale | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Balance
Change in Modified Aschworth scale | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Spasticity
Change in 2 minutes walk test | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Walking
Change in Alberts test | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Neglect
Change in EQ5D | Assessed at baseline, after 4 weeks of training and 6 months after stroke
  Health outcome
Stroke impact scale | 6 months after stroke
  Functioning and disability

CONTACTS AND LOCATIONS:
Overall Officials: Jörgen Borg, Professor, Principal Investigator — Department of Rehabilitation medicine, Danderyd Hospital, Karolinska Institute
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County, Sweden

REFERENCES:
- [Background] Nilsson A, Vreede KS, Haglund V, Kawamoto H, Sankai Y, Borg J. Gait training early after stroke with a new exoskeleton--the hybrid assistive limb: a study of safety and feasibility. J Neuroeng Rehabil. 2014 Jun 2;11:92. doi: 10.1186/1743-0003-11-92. PMID 24890413
- [Derived] Wall A, Palmcrantz S, Borg J, Gutierrez-Farewik EM. Gait pattern after electromechanically-assisted gait training with the Hybrid Assistive Limb and conventional gait training in sub-acute stroke rehabilitation-A subsample from a randomized controlled trial. Front Neurol. 2023 Oct 11;14:1244287. doi: 10.3389/fneur.2023.1244287. eCollection 2023. PMID 37885482